CLINICAL TRIAL: NCT03987282
Title: Implementation of Seek, Test, Treat & Retain Strategies Among People Who Inject Drugs in Malaysia
Brief Title: Implementation of STTR Strategies Among People Who Inject Drugs in Malaysia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial on hold
Sponsor: Yale University (Other)
Collaborators: Universiti Sains Malaysia (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2000023790; 1R01DA047789-01 (NIH)
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: HIV Seropositivity; Opioid-use Disorder
MeSH Terms: conditions — HIV Seropositivity; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Pre- versus post-implementation evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care (EUC) (Active Comparator): The EUC consists of provision of ART and medical care for HIV and other medical HIV co-morbidities provided at the HIV/AIDS treatment center with an expedited and facilitated referral to a methadone maintenance treatment (MMT).
  Interventions: Other: Enhanced usual care (EUC)
- Fully Implemented Seek-Test-Treat-Retain (FI-STTR) model (Experimental): The FI-STTR care model will include the usual care supplemented by continuing education and coaching of medical staff at HIV/AIDS and MMT clinics and by provision of additional peer-based counseling intervention
  Interventions: Other: Enhanced usual care (EUC); Behavioral: Peer-based counseling

INTERVENTIONS:
Other: Enhanced usual care (EUC) — Provision of ART and medical care for HIV and other medical HIV co-morbidities provided at the HIV/AIDS treatment center with an expedited and facilitated referral to a methadone maintenance treatment (MMT).
Behavioral: Peer-based counseling — Peer-based counseling intervention focused on behavioral skills and strategies that patients can learn and master to achieve uninterrupted, long-term ART treatment participation while continuing OUD recovery through MMT
  Arms: Fully Implemented Seek-Test-Treat-Retain (FI-STTR) model

SUMMARY:
This pragmatic, multisite, implementation and effectiveness research evaluates a strategy to improve HIV treatment outcomes (increased rates of patients on ART with virological suppression, improved treatment retention and ART adherence) for people living with HIV (PLWH) with opioid use disorder (OUD). Engaging 4 large regional HIV/AIDS treatment centers in Malaysia, the study will evaluate barriers and facilitators for implementation of improved care model and will evaluate the comparative effectiveness of the model in a clinical trial. The research will provide critically important evidence for implementation of effective Seek-Test-Treat, and Retain models for PLWH and OUD throughout Malaysia and inform healthcare policy in other low to middle income countries and regions with limited healthcare resources.

DETAILED DESCRIPTION:
At each of the study locations, individuals testing HIV positive who also have OUD (n=4x70) will receive concurrent anti-retroviral therapy (ART) and methadone maintenance treatment (MMT) based on the usual care standards. Their patient level outcomes will be compared with individuals meeting the same inclusion criteria (n=4x70) and treated under the proposed improved model (post implementation evaluation). The usual care standard will consist of provision of ART and medical care for HIV and other medical HIV co-morbidities provided at the HIV/AIDS treatment center with an expedited and facilitated referral to a methadone maintenance treatment (MMT). The improved care model will include the usual care supplemented by continuing education and coaching of medical staff at HIV/AIDS and MMT clinics and by provision of additional peer-based counseling intervention focused on behavioral skills and strategies that patients can learn and master to achieve uninterrupted, long-term ART treatment participation while continuing OUD recovery through MMT. The primary outcome measure, rates of patients with virologic suppression (< 20 copies/mL) in the two care models will be assessed at 24 weeks. The secondary outcomes, also followed for 24 weeks, will include ART adherence measured by objective measures (tenofovir dried blood spots, clinic records) and self-report; decreased illicit opioid use measured by rates of opioid negative urine toxicology results and self-report; and improvements on other health-related and functional status outcomes.

Aim 1: To evaluate comparative effectiveness of fully implemented seek, test, treat and retain strategy (FI-STTR) the study will compare clinical, patient level, outcomes between enhanced usual care (EUC) and FI-STTR across the four study sites.

Hypothesis: The investigators hypothesize a statistically significant effect on the primary outcome favoring the FI-STTR over EUC. It is also hypothesized that FI-STTR will be superior over EUC on all secondary outcomes.

Concurrently at each study location, using implementation science mixed methods research tools and engaging key local stakeholders (treatment providers, patients, their families, and community activists), and evaluating clinical and healthcare data, the study will assess existing barriers (organizational, personnel, and community level factors) and uncover available resources and facilitators for a successful implementation of the improved care model.

Aim 2: To assess existing barriers; organizational, personnel, community level factors; and available resources and potentially facilitating factors for successful implementation of the FI-STTR at HIV/AIDS clinics. There are no hypotheses specified a priori for Aim 2 of the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* potential participants must meet the inclusion criteria for ART and MMT and begin receiving these treatments

Exclusion Criteria:

* ART and MMT exclusion criteria include: liver enzymes greater than 5 times the upper limit of normal (ULN); liver failure (Childs Pugh Turcot Grade B or C).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 560 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Virologic suppression | 24 weeks
  The rates of patients with virologic suppression (< 20 copies/mL) in the two care models will be assessed at 24 weeks

SECONDARY OUTCOMES:
ART adherence, proportion of days when medication is taken as prescribed | 24 weeks
  ART adherence will be assessed by self-report using a timeline follow back (TLFB) methodology
Opioid use | 24 weeks
  Illicit opioid use measured by rates of opioid negative urine toxicology results and self-report
Depression scores | 24 weeks
  Center for Epidemiological Studies Depression Scale (CES-D) total score. The scale range is from 0 to 60; higher scores indicate more depression symptoms.
Psychiatric symptoms | 24 weeks
  Brief Symptom Inventory (BSI) a 53-item self-report inventory in which participants rate the extent to which they have been bothered (0 ="not at all" to 4="extremely") in the past week by various symptoms. The BSI has nine subscales designed to assess individual symptom groups: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. Higher scores indicate higher severity of symptoms.
Changes in the quality of life index | 24 weeks
  Short version of the World Health Organization Quality of Life (WHOQOL-BREF). The WHOQOL-BREF contains a total of 26 questions. In addition, two items from the Overall quality of Life and General Health facet are included. Four domains are assessed: Physical, Psychological, Social Relationship, and Environment.

CONTACTS AND LOCATIONS:
Overall Officials: Marek C Chawarski, PhD, Principal Investigator — Yale University
Locations (1):
- Universiti Sains Malalysia, Tasek Gelugor, Pulau Pinang, Malaysia